CLINICAL TRIAL: NCT04180423
Title: What Factors Affect Operating Room Efficiency When Performing TKA Using Customized Implant Techniques: Conformis iTotal (CR), (PS)
Brief Title: TKA Operating Room Efficiency for TKA Using Customized Implant Techniques
Status: Terminated | Type: Observational
Why Stopped: Decision of investigational team
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-002i
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Off-the-Shelf Total Knee Arthroplasty Patients
  Interventions: Device: Off-the-Shelf Implant Total Knee Replacement
- Conformis iTotal Total Knee Arthroplasty Patients
  Interventions: Device: Customized Implant Total Knee Replacement

INTERVENTIONS:
Device: Off-the-Shelf Implant Total Knee Replacement — Total Knee Replacement, or knee arthroplasty, is a common surgical procedure performed to relieve the pain and disability resulting from osteoarthritis. In general, the surgery consists of replacing the diseased or damaged joint surfaces of the knee with metal and plastic components shaped to allow continued motion of the knee. Off-the-Shelf implants use standard sizing.
  Groups: Off-the-Shelf Total Knee Arthroplasty Patients
Device: Customized Implant Total Knee Replacement — Total Knee Replacement, or knee arthroplasty, is a common surgical procedure performed to relieve the pain and disability resulting from osteoarthritis. In general, the surgery consists of replacing the diseased or damaged joint surfaces of the knee with metal and plastic components shaped to allow continued motion of the knee. Customized implants are customized individually made knee implants which are designed specific to each patient's unique anatomy.
  Other Names: Conformis iTotal
  Groups: Conformis iTotal Total Knee Arthroplasty Patients

SUMMARY:
This is a multi-centered prospective, consecutively enrolled study that will be conducted in the United States. Surgeons that are new users of the iTotal Knee system (defined by no experience using the customized Total Knee Replacement (TKR) in the last 6 months) will be involved in the study. To complete the study protocol, the center will collect baseline surgical and training data on 10 "off-the-shelf" TKR patients using the implant system the surgeon currently uses. Then the first 50 consecutive patients who have been identified to receive the iTotal implant (Cruciate-Retaining or Posterior-Stabilizing) based on patient factors and the implant system IFU will be enrolled in the study. Simultaneous bilateral Total Knee Arthroplasty cases will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age

Exclusion Criteria:

* Participation in another clinical study which would confound results
* Inability to complete the protocol in the opinion of the clinical staff due to safety or other reasons
* Simultaneous bilateral Total Knee Arthroplasty cases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving Total Knee Arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Operating Room Efficiency | Single time point - day of surgery
  Surgeon questionnaire to determine operating room efficiency from the 1st to the 50th iTotal implant performed and to determine any differences that might exist between operating room efficiency between the iTotal surgery and baseline metrics when performing OTS implant surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Kettering Medical Center, Kettering, Ohio, United States

IPD SHARING:
Plan to Share IPD: No